CLINICAL TRIAL: NCT00246090
Title: A Phase II Open Label Single-Arm Study of E7389 in Patients With Locally Advanced or Metastatic Breast Cancer, Previously Treated With Anthracycline, Taxane, and Capecitabine Therapy, Refractory to the Last Prior Therapy for Their Disease
Brief Title: A Phase II Study of E7389 in Patients With Breast Cancer, Previously Treated With Anthracycline, Taxane and Capecitabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Eisai Limited (Industry)
Responsible Party: Eisai Medical Services, Eisai Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-G000-211; 2005-003656-35 (EudraCT Number)
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E7389

INTERVENTIONS:
Drug: E7389 — E7389 1.4 mg/m^2 intravenous bolus given over 2-5 minutes on Days 1 and 8 every 21 days.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of E7389 in Patients with locally advanced or metastatic breast cancer, previously treated with anthracycline, taxane, and capecitabine as prior therapy, and who are refractory to the last prior therapy for their disease.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with histologically or cytologically confirmed carcinoma of the breast. Every effort should be made to make paraffin embedded tissue or slides from the diagnostic biopsy or surgical specimen available for confirmation of diagnosis.
2. Patients with locally advanced or metastatic disease who have received at least two (and not more than five) prior chemotherapeutic regimens for breast cancer, at least one of which was administered for treatment of locally advanced or metastatic disease.

   Prior therapy must be documented by the following criteria prior to entry onto study:
   * Regimens must have included an anthracycline (eg, doxorubicin, epirubicin), a taxane (eg, paclitaxel, docetaxel) and capecitabine in any combination or order.
   * One or two of these regimens may have been administered as adjuvant and/or neoadjuvant therapy.
   * Patients with human epidermal growth factor receptor 2 (HER2/neu) over-expressing tumors must additionally have been treated with trastuzumab.
   * Patients with estrogen receptor-expressing tumors may have additionally been treated with estrogen-specific therapy.
   * Prior hormonal therapy, biological therapy, (eg, trastuzumab, bevacizumab), or immunotherapy, is not to be counted as one of the 2 to 5 prior chemotherapy regimens allowed. However, hormonal therapy must be discontinued one week before administration of E7389, and biological therapy must be discontinued two weeks before E7389 administration.
   * Patients who are being treated with bisphosphonates when they enter the study are allowed to continue the medication as long as the dosing does not change. In case a change in dosing is deemed necessary, the case needs to be discussed with the Sponsor.
3. Progression on or within six months of the last regimen for advanced disease, documented by the following:

   * The dates of treatment, doses, outcome of therapy and the reason for discontinuation of prior anthracycline, taxane, capecitabine, and trastuzumab therapy must be provided.
   * Prior to entry onto the study, information ensuring that the last therapy fulfills eligibility criteria is required, which includes progression while receiving this last prior chemotherapy regimen, or within six months of receiving that therapy.
   * Chemotherapy medication administration sheets or other official medical/hospital records indicating type and dates of chemotherapy must be available for inspection, and one of the following as a reason for discontinuation of medication is required: radiographic evidence of progression, or doctor's office or hospitalization notes documenting radiologic progression, clinically documented increase in tumor burden, and/or increase in tumor-specific markers.
4. Patients with measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, defined as at least one lesion that can be accurately measured in at least one diameter (at least 10 mm in longest diameter [LD] by spiral computer tomography [CT] scan), or at least 20 mm by standard techniques. If the only measurable lesion is a lymph node, it must measure at least 20 mm in LD. If a single lesion is identified as the target lesion, a biopsy or aspiration with cytological or histological confirmation of the diagnosis of breast carcinoma is required.
5. Resolution of all chemotherapy or radiation-related toxicities to less than Grade 2 severity, except for stable sensory neuropathy ≤ Grade 2 and alopecia.
6. Age >= 18 years.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
8. Life expectancy of ≥ 3 months.
9. Adequate renal function as evidenced by serum creatinine ≤ 2.0 mg/dL or calculated creatinine clearance ≥ 40 mL/minute (min) per the Cockcroft and Gault formula.
10. Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) ≥1.5 x 10^9/L hemoglobin ≥ 10.0 g/dL (acceptable if it is corrected by therapeutic intervention or transfusional support), and platelet count ≥ 100 x 10^9/L.
11. Adequate liver function as evidenced by bilirubin ≤ 1.5 mg/dL and alkaline phosphatase, alanine transaminase (ALT), and aspartate transaminase (AST) ≤ 3 times the upper limits of normal (ULN) (in the case of liver metastases ≤ 5 x ULN), unless there are bone metastases, in which case liver specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of the total alkaline phosphatase.
12. Willing and able to complete the European Organization for Research on the Treatment of Cancer (EORTC) quality of life assessment, Analgesic Diary, and Pain Visual Analog Scale (VAS).
13. Willing and able to comply with the study protocol for the duration of the study.
14. Written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

Exclusion Criteria:

1. Patients must not have received chemotherapy, radiation, or biologic therapy within two weeks, hormonal therapy within one week, or trastuzumab within three weeks, before E7389 treatment start.
2. Patients must not have received radiation therapy encompassing > 30% of marrow (a lesion that has been irradiated cannot be used as a target lesion, unless it has progressed after the irradiation).
3. Patients must not have pre-existing neuropathy > Grade 2.
4. Patients must not have participated in a prior E7389 clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2005-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dale Shuster, Ph.D., Study Director — Eisai Inc.
Locations (63):
- United States (58):
  - Birmingham Hematology and Oncology, Birmingham, Alabama
  - Mercy Cancer Center, Hot Springs, Arkansas
  - Arkansas Cancer Research Center, Little Rock, Arkansas
  - Wilshire Oncology Medical Group, Inc., La Verne, California
  - Rocky Mountain Cancer Center-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Center-Rose, Denver, Colorado
  - Rocky Mountain Cancer Center, Littleton, Colorado
  - Cancer Research Network, Plantation, Florida
  - Hematology-Oncology Associates, Port Saint Lucie, Florida
  - Dr. Elizabeth Tan-Chiu, PA, Tamarac, Florida
  - Peachtree Hematology And Oncology Consultants, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Cancer Care and Hematology Specialist of Chicagoland, Niles, Illinois
  - Central Indiana Cancer Center, Indianapolis, Indiana
  - Monroe Medical Center, Munster, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Frederick Memorial Hospital, Regional Cancer Therapy Center, Frederick, Maryland
  - Park Nicollet Institute, Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Montana Cancer Specialists, Missoula, Montana
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - New York Oncology Hematology, P.C, Albany, New York
  - North Shore Hematology Oncology Associates, East Setakuet, New York
  - Huntington Medical Group, PC, Huntington Station, New York
  - Weill Cornell Breast Cancer Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Northwestern Carolina Oncology And Hematology, PA, Hudson, North Carolina
  - Raleigh Hematology Oncology Associates, Raleigh, North Carolina
  - 'Signal Point Hematology/Oncology, Inc., Middletown, Ohio
  - Medical University of Ohio, Toledo, Ohio
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Northwest Cancer Specialist Rose Qtr, Portland, Oregon
  - Kaiser Permanente, Central Interstate Clinic, Hematology Oncology, Portland, Oregon
  - Northwest Cancer Specialist Hoyt, Portland, Oregon
  - Charleston Hematology Oncology, Charleston, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Texas Oncology, P.A. Bedford, Bedford, Texas
  - Center For Oncology Research and Treatment, PA, Dallas, Texas
  - Texas Oncology PA, Dallas, Texas
  - Sammons Cancer Center-Dallas, Dallas, Texas
  - El Paso Cancer Treatment Center West, El Paso, Texas
  - El Paso Cancer Treatment Center, El Paso, Texas
  - Texas Oncology PA, Houston, Texas
  - Baylor College of Medicine, Breast Cancer Clinic, Houston, Texas
  - North Texas Regional Cancer Center, Plano, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Valley Oncology PA, Weslaco, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Fairfax Northern VA Hematology Oncology PC, Fairfax, Virginia
  - Oncology and Hematology Associates, Salem, Virginia
  - Cancer Care Northwest, Spokane, Washington
  - Northwest Cancer Specialist, Vancouver, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
- Canada (5):
  - Hamilton Health Sciences Juravinski Cancer Centre, Hamilton, Ontario
  - NW Ontario Regional Cancer Centre, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Centre Hospitaliere Universitaire de Montreal, Montreal, Quebec
  - McGill University, Dept. of Oncology, Clinical Research Program, Montreal, Quebec

REFERENCES:
- [Derived] Muss H, Cortes J, Vahdat LT, Cardoso F, Twelves C, Wanders J, Dutcus CE, Yang J, Seegobin S, O'Shaughnessy J. Eribulin monotherapy in patients aged 70 years and older with metastatic breast cancer. Oncologist. 2014 Apr;19(4):318-27. doi: 10.1634/theoncologist.2013-0282. Epub 2014 Mar 28. PMID 24682463

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 42 centers in US and 36 centers in EU during the period of Oct 2005 to Sep 2007.
Groups:
- E7389 1.4 mg/m^2: E7389 1.4 mg/m^2 intravenous bolus given over 2-5 minutes on Days 1 and 8 every 21 days.
Period: Overall Study
Arm/Group | E7389 1.4 mg/m^2
Started | 298
Completed | 3
Not Completed | 295
Not completed — Adverse Event | 25
Not completed — Withdrawal by Subject | 7
Not completed — Progressive Disease | 212
Not completed — Clinical Progression | 30
Not completed — Physician Decision | 11
Not completed — Not Otherwise Specified | 10

BASELINE CHARACTERISTICS:
Arm/Group | E7389 1.4 mg/m^2
Number analyzed (Participants) | 291
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety Population
  years | 55.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 291
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian/Pacific Islander | 6
  Black or African American | 12
  White | 199
  Other | 8
  Unknown or Not Reported | 66

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Based on Response Evaluation Criteria in Solid Tumors (RECIST), consisting of complete response (CR) plus partial response (PR). Defined as the best response from the start of treatment until disease progression or recurrence. Lesions measured by computed tomography (CT) scan and magnetic resonance imaging (MRI). Objective response rate: complete response (CR-disappearance of all lesions)+ partial response (PR-30% decrease in lesion diameter), Progressive Disease (PD-20% increase in lesion diameter), stable disease (SD-neither shrinkage nor increase of lesions).
Time Frame: Every two cycles
Population: Eligible Population
Measure: Number; unit: Percentage of Participants
Arm/Group | E7389 1.4 mg/m^2
Number analyzed (Participants) | 269
Percentage of Participants | 14.1

2. Secondary Outcome: Duration of Response
Description: Complete response (CR) is defined as the disappearance of all lesions. Partial response (PR) is defined as 30% decrease in lesion diameter.
Time Frame: From first documented complete or partial response until disease progression or death
Population: Eligible Population
Measure: Median (Full Range); unit: Days
Arm/Group | E7389 1.4 mg/m^2
Number analyzed (Participants) | 38
Days | 176 [29 to 258]

ADVERSE EVENTS:
Arm/Group | E7389 1.4 mg/m^2
Serious Adverse Events (participants affected / at risk) | 88/291
Other Adverse Events (participants affected / at risk) | 290/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 1.4 mg/m^2 (N=291)
Anemia (Blood and lymphatic system disorders) | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Cardiac Arrest (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Diplopia (Eye disorders) | 1
Macular Hole (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 2
Chest Pain (General disorders) | 1
Death (General disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 4
Pyrexia (General disorders) | 11
Biliary Dilatation (Hepatobiliary disorders) | 1
Bacteremia (Infections and infestations) | 1
Bacterial Sepsis (Infections and infestations) | 1
Clostridium Difficile Colitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Neutropenic Infection (Infections and infestations) | 1
Neutropenic Sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Septic Shock (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypovolemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Lymphangiosis Carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to Central Nervous (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to Retroperitoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 1
Spinal Cord Compression (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Confusional State (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Mental Status Changes (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 7
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 1.4 mg/m^2 (N=291)
Anemia (Blood and lymphatic system disorders) | 86
Febrile Neutropenia (Blood and lymphatic system disorders) | 16
Leukopenia (Blood and lymphatic system disorders) | 64
Neutropenia (Blood and lymphatic system disorders) | 174
Lacrimation Increased (Eye disorders) | 31
Abdominal Distention (Gastrointestinal disorders) | 16
Abdominal Pain (Gastrointestinal disorders) | 38
Abdominal Pain Upper (Gastrointestinal disorders) | 26
Constipation (Gastrointestinal disorders) | 96
Diarrhea (Gastrointestinal disorders) | 65
Dry Mouth (Gastrointestinal disorders) | 25
Dyspepsia (Gastrointestinal disorders) | 27
Nausea (Gastrointestinal disorders) | 141
Stomatitis (Gastrointestinal disorders) | 32
Vomiting (Gastrointestinal disorders) | 72
Asthenia (General disorders) | 112
Chest Pain (General disorders) | 24
Fatigue (General disorders) | 107
Mucosal Inflammation (General disorders) | 44
Peripheral Edema (General disorders) | 37
Pain (General disorders) | 32
Pyrexia (General disorders) | 88
Urinary Tract Infection (Infections and infestations) | 35
Weight Decreased (Investigations) | 29
Anorexia (Metabolism and nutrition disorders) | 74
Hypokalemia (Metabolism and nutrition disorders) | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 48
Back Pain (Musculoskeletal and connective tissue disorders) | 46
Bone Pain (Musculoskeletal and connective tissue disorders) | 30
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 17
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 16
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 20
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 30
Myalgia (Musculoskeletal and connective tissue disorders) | 42
Neck Pain (Musculoskeletal and connective tissue disorders) | 17
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 38
Dizziness (Nervous system disorders) | 28
Dysgeusia (Nervous system disorders) | 40
Headache (Nervous system disorders) | 61
Neuropathy (Nervous system disorders) | 24
Neuropathy Peripheral (Nervous system disorders) | 30
Paraesthesia (Nervous system disorders) | 33
Peripheral Sensory Neuropathy (Nervous system disorders) | 28
Anxiety (Psychiatric disorders) | 27
Depression (Psychiatric disorders) | 26
Insomnia (Psychiatric disorders) | 33
Cough (Respiratory, thoracic and mediastinal disorders) | 57
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 57
Pharyngolarygeal Pain (Respiratory, thoracic and mediastinal disorders) | 20
Alopecia (Skin and subcutaneous tissue disorders) | 179
Rash (Skin and subcutaneous tissue disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No